CLINICAL TRIAL: NCT04004871
Title: The Efficacy and Safety of Induction Chemotherapy With Nab-paclitaxel, Cisplatin and Fluorouracil, Concurrent Chemotherapy of Cisplatin and IMRT in Locoregionally Advanced Nasopharyngeal Carcinoma: A Prospective, Multi-centeric, Open, Non-controlled, Phase II Clinical Trial
Brief Title: Induction Chemotherapy With Nab-paclitaxel, Cisplatin and Fluorouracil for Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Collaborators: Liuzhou Workers' Hospital (Other Government); Wuzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kai Hu, Clinical Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMUHK1
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer; Nasopharynx Cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Fluorouracil; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction chemotherapy and concurrent chemoradiotherapy (Experimental): Patients receive induction chemotherapy with Nab-paclitaxel, cisplatin and fluorouracil every three weeks for three cycles before radiotherapy, and then receive concurrent chemoradiotherapy.
  Interventions: Drug: Nab-paclitaxel, Cisplatin and Fluorouracil; Radiation: concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Nab-paclitaxel, Cisplatin and Fluorouracil — Patients receive Nab-paclitaxel (200mg/m2 on day 1), cisplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before concurrent chemoradiotherapy.
  Other Names: APF induction chemotherapy
Radiation: concurrent chemoradiotherapy — Patients receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Other Names: Radical radiotherapy and concurrent cisplatin

SUMMARY:
Nasopharyngeal carcinoma (NPC) is commonly observed in southern China, particularly in the Pearl River delta area and the Xijiang River basin in the Guangdong and Guangxi provinces, with an incidence rate as high as 25-50 per 100,000. The National Comprehensive Cancer Network guidelines (version 1, 2018), have recommended use of induction chemotherapy followed by CCRT as category 2A for NPC, especially the TPF regimen as category 1 for EBV-associated disease. The nanoparticle albumin-bound paclitaxel (Nab-paclitaxel) is a promising new agent with more efficient entry to the tumor microenvironment and preferential uptake by cancer cells. Superior activity of Nab-paclitaxel regimens without the necessity for antianaphylactic pretreatments has been shown in various solid tumors compared with the traditional solvent-based paclitaxel-based ones. However, the safety and efficacy of combination of Nab-paclitaxel, cisplatin and Fluorouracil (APF) has not been determined in patients with locoregionally advanced NPC. In this prospective, Multi-centeric, Open, Non-controlled phase II clinical trial, investigators perform an exploratory study to the efficacy and Safety of APF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
2. Tumor staged as T3-4/N1-3 (according to the 8th UICC edition).
3. No evidence of distant metastasis (M0).
4. EBV positive.
5. Satisfactory performance status: ECOG≤2.
6. Adequate marrow: leucocyte count ≥4000/uL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
7. Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
8. Adequate renal function: creatinine clearance ≥60 ml/min.
9. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
2. Age>60 years or <18 years.
3. Treatment with palliative intent.
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
5. Pregnancy or lactation.
6. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
7. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  To be determined by measurement of target lesions according to RECIST criteria

SECONDARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  From the date of registration to the date of either locally, regionally or distant failure or last follow-up
Overall survival（OS） | 3 years
  From the date of registration to the date of death is observed or to last follow-up visit
Adverse Events | 3 years
  Incidence of Treatment-Emergent Adverse Events Evaluated according to NCI-CTC AE V4.03

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China